CLINICAL TRIAL: NCT06259240
Title: Prone Plank Exercises Versus Electrical Stimulation in Treatment of Diastasis Rectus Abdominis in Postpartum Women
Brief Title: Prone Plank Exercises for Diastasis Rectus Abdominis in Postpartum Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rowida Abd Elgleel Sayed Abd Elgleel, Senior at Outpatient Clinics, Faculty of Physical Therapy, Cairo University., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Plank Exercises in Diastasis
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Post Partum Women
MeSH Terms: interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone Plank Exercises (Active Comparator): Forty two post partum woman will recieve progressive prone plank exercises, three times a week, for eight weeks, and with a moderate hard intensity.
  Interventions: Other: Prone plank exercises
- Electrical Stimulation (Sham Comparator): Forty two post partum woman will recieve electrical stimulation for the rectus abdominis muscle day after day for 8 weeks. The patient position was relaxed in the crook lying position. The session parameters were 30 minutes/session with a low frequency current (50-100Hz).
  Interventions: Device: Electrical Stimulation

INTERVENTIONS:
Other: Prone plank exercises — Patients in this group will recieve prone plank exercises, three times a week, for eight weeks, and with a moderate hard intensity. During the first four weeks, the exercises session began with light walking for five minutes followed by corrected exercises. Firstly, women will perform stable prone plank exercises. Secondly, women will be asked to apply the unilateral position of prone plank. Thirdly, using a 65 cm diameter Swiss ball, women will be asked to assume the prone bridge position. During the last four weeks, women will be asked to repeat the same program noting that the progressive prone plank exercises should be applied in a dosage of 20 repetitions, three sets, holding the contraction for one minute, and taking a break for two minutes.
  Arms: Prone Plank Exercises
Device: Electrical Stimulation — Electrical Stimulation
  Arms: Electrical Stimulation

SUMMARY:
The purpose of this study was to compare between the effects of prone plank exercises versus ES for DRA in postpartum women.

DETAILED DESCRIPTION:
The study conducted on forty-two woman. They had diastasis rectus abdominis12 weeks to 36 months postpartum. They were randomly divided into two equal groups; group A received prone plank exercises while group B recieved electrical stimulation.All patients recieved three sessions per week foe eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* they had DRA 12 weeks to 36 months postpartum, and were referred to physiotherapy by a gynaecologist, multiparous with the IRD measuring greater than two cm. Age ranged between 20-35 years. Body mass index didn't exceed 30 kg/m2.

Exclusion Criteria:

* they were in ongoing pregnancy, twin pregnancy, premature birth before gestation week 37, and exceeded more than thirty-six months postpartum.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 42 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Imaging Device | Eight weeks after the beginning of the intervention
  Changes in Interrectus distance above umbilicus at rest from baseline to four weeks after the beginning of intervention
Ultrasound Imaging Device | Eight weeks after the beginning of the intervention
  Changes in Interrectus distance below umblicus at rest from baseline to four weeks after the beginning of intervention
Ultrasound Imaging Device | Eight weeks after the beginning of the intervention
  Changes in Interrectus distance above umbilicus at contraction from baseline to four weeks after the beginning of intervention
Ultrasound Imaging Device | Eight weeks after the beginning of the intervention
  Changes in Interrectus distance below umbilicus at contractionfrom baseline to four weeks after the beginning of intervention

SECONDARY OUTCOMES:
The measuring tape | Eight weeks after the beginning of the intervention
  Changes in waist hip ratio from baseline to four weeks after the beginning of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Fayiz Elshamy, Professor, Study Director — Kafrelsheikh University
Locations (1):
- Faculty of physical therapy labs at kafr El sheikh University, Kafr ash Shaykh, Egypt